CLINICAL TRIAL: NCT02698280
Title: Phase II Study of Bevacizumab and Nimustine in Patients With Recurrent High Grade Glioma
Brief Title: Bevacizumab and Nimustine in Patients With Recurrent High Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiaojie Ding, Resident, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2015-289; 02
Record Dates: First submitted 2016-02-20; First posted 2016-03-03 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Glioblastoma
Keywords: Bevacizumab; Nimustine; Pathology, Molecular
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Nimustine

ARMS (1):
- Treatment (Experimental): Patients are treated with bevacizumab and nimustine. Every 6 weeks is defined as one therapeutic cycle. Adverse effect is evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE; version 4.03). Hematologic toxicity is evaluated every 2 weeks. Liver function, renal function, and electrolytes are assessed every 4-6 weeks. Platelet should be no less than 100*10^9/L and neutrophil count should be no less than 1.5*10^9/L.
  Interventions: Drug: Bevacizumab; Drug: Nimustine

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is administered intravenously at 5mg/kg every 3 weeks.
  Other Names: Avastin
Drug: Nimustine — Nimustine is administered intravenously at 90mg/m^2 to 110mg/m^2 every 6 weeks.

SUMMARY:
The purpose of this study is to determine whether bevacizumab and nimustine are effective in the treatment of recurrent high grade glioma and to explore whether there is any subgroup being sensitive to this therapeutic protocol.

DETAILED DESCRIPTION:
Although anti-angiogenesis therapy for glioblastoma(GBM) are showing promise, GBMs often develop resistance to treatment within months or weeks after salvage therapy. There are still no effective markers to predict the response rate to bevacizumab.

So the investigators initiate a single-arm Phase II study to evaluate the efficacy and tolerability of bevacizumab and nimustine regimen and to explore the predictive markers in patients with recurrent high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary tumor as high-grade gliomas (WHO III or IV)
* All patients should complete radiotherapy and chemotherapy for primary gliomas
* Enhanced MRI and magnetic resonance spectroscopy showed unequivocal evidence of tumor recurrence or progression.
* Those patients underwent surgical resection after tumor recurrence can also be enrolled if histological diagnosis of GBM is available, and MRI within 3 days after operation is needed.
* The patients with recurrent gliomas didn't undergo bevacizumab therapy before enrollment.
* The time to be enrolled should be more than 90 days after the radiation therapy, more than 28 days after operation for recurrent tumor or prior chemotherapy.
* Eastern Cooperative Oncology Group score: 0-2
* Written informed consent
* Laboratory test: Neutrophil count > 1.5*10^9/L, platelet count > 100*109/L, hemoglobin > 8 g/dL, blood urea nitrogen and creatinine < 1.5 upper limit of normal(ULN), blood total bilirubin and conjugated bilirubin < 1.5 ULN, alanine aminotransferase(ALT) and aspartate aminotransferase(AST) < 3 ULN, alkaline phosphatase(AKP) < 2 ULN

Exclusion Criteria:

* Pregnant or lactating women
* Allergic to administered drugs
* Radiation therapy in the previous 90 days before enrollment
* The patients with recurrent gliomas were treated with bevacizumab therapy before enrollment.
* Acute infection in need of antibiotics intravenously
* Participation in other clinical trials in the 90 days before enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
All cause response to treatment | 3 weeks
  Response will be evaluated according to the Response Assessment in Neuro-Oncology(RANO) criteria.Imaging Data (postcontrast T1W,T2/FLAIR),clinical symptoms and corticosteroid use will be collected in each participant and response assessment will be performed by one neurosurgeon and one neuroradiologist.

SECONDARY OUTCOMES:
All cause mortality | One year
All cause disease progression | 3 weeks
  Progression disease will be evaluated according to the RANO criteria
All cause severe toxicities | 3 weeks
  All toxicities will be assessed and graded according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Yu Yao, MD, PhD, Study Chair — Department of Neurosurgery, Huashan hospital; Daoying Geng, MD, Study Chair — Department of Radiology, Huashan hospital; Xiaojie Ding, MD, Principal Investigator — Department of Neurosurgery, Huashan hospital; Jianbo Wen, MD, Principal Investigator — Department of Radiology, Huashan hospital
Locations (1):
- Huashan hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Vredenburgh JJ, Desjardins A, Reardon DA, Friedman HS. Experience with irinotecan for the treatment of malignant glioma. Neuro Oncol. 2009 Feb;11(1):80-91. doi: 10.1215/15228517-2008-075. Epub 2008 Sep 10. PMID 18784279
- [Background] Reardon DA, Wen PY, Desjardins A, Batchelor TT, Vredenburgh JJ. Glioblastoma multiforme: an emerging paradigm of anti-VEGF therapy. Expert Opin Biol Ther. 2008 Apr;8(4):541-53. doi: 10.1517/14712598.8.4.541. PMID 18352856
- [Background] Taal W, Oosterkamp HM, Walenkamp AM, Dubbink HJ, Beerepoot LV, Hanse MC, Buter J, Honkoop AH, Boerman D, de Vos FY, Dinjens WN, Enting RH, Taphoorn MJ, van den Berkmortel FW, Jansen RL, Brandsma D, Bromberg JE, van Heuvel I, Vernhout RM, van der Holt B, van den Bent MJ. Single-agent bevacizumab or lomustine versus a combination of bevacizumab plus lomustine in patients with recurrent glioblastoma (BELOB trial): a randomised controlled phase 2 trial. Lancet Oncol. 2014 Aug;15(9):943-53. doi: 10.1016/S1470-2045(14)70314-6. Epub 2014 Jul 15. PMID 25035291
- [Background] Killela PJ, Pirozzi CJ, Healy P, Reitman ZJ, Lipp E, Rasheed BA, Yang R, Diplas BH, Wang Z, Greer PK, Zhu H, Wang CY, Carpenter AB, Friedman H, Friedman AH, Keir ST, He J, He Y, McLendon RE, Herndon JE 2nd, Yan H, Bigner DD. Mutations in IDH1, IDH2, and in the TERT promoter define clinically distinct subgroups of adult malignant gliomas. Oncotarget. 2014 Mar 30;5(6):1515-25. doi: 10.18632/oncotarget.1765. PMID 24722048
- [Background] Chan AK, Yao Y, Zhang Z, Chung NY, Liu JS, Li KK, Shi Z, Chan DT, Poon WS, Zhou L, Ng HK. TERT promoter mutations contribute to subset prognostication of lower-grade gliomas. Mod Pathol. 2015 Feb;28(2):177-86. doi: 10.1038/modpathol.2014.94. Epub 2014 Aug 1. PMID 25081751